CLINICAL TRIAL: NCT00476034
Title: A 39-week, Double-blind, Active-controlled Extension to CCOX189A2361, a 13-week, Multicenter, Randomized, Double-blind, Double-dummy, Placebo-controlled, Parallel Trial of 2 Different Dose Regimens of Lumiracoxib (100 mg od and 200 mg od Initial Dose for Two Weeks Followed by 100 mg od) in Patients With Primary Knee Osteoarthritis, Using Celecoxib (200 mg od) as a Comparator
Brief Title: Efficacy and Safety of Lumiracoxib in Patients With Primary Knee Osteoarthritis (OA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCOX189A2361E1
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; lumiracoxib; celecoxib; Cox-2; knee
MeSH Terms: conditions — Osteoarthritis | interventions — lumiracoxib

INTERVENTIONS:
Drug: lumiracoxib

SUMMARY:
This 39-week, active controlled, study is designed to assess long-term efficacy, safety and tolerability of lumiracoxib 100mg od in patients with osteoarthritis (OA) of the knee who participated in the 13-week core CCOX189A2361 study.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who completed the core study 2361 may enter the extension trial upon signing informed consent. A patient is defined as completing if he/she completed the core study 2361 up to and including Visit 6 (week 13) without a major protocol violation.

Exclusion Criteria:

* Those patients for whom continued treatment in the extension study is not considered appropriate by the treating physician
* Those patients who were non-compliant or who demonstrated a major protocol violation in the core study.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 1312 (Actual)
Dates: Start 2003-12; Primary Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
To compare lumiracoxib 100mg od to celecoxib 200mg od in treating osteoarthritis (OS) of the target knee with respect to:
Overall OA pain intensity in the target knee on a 0-100 mm Visual Analog Scale (VAS) at 26 weeks.
Patient's global assessment of disease activity on a 0-100mm VAS at 26 weeks.
Patient's functional status using the WOMAC total score at 26 weeks

SECONDARY OUTCOMES:
To assess the safety and tolerability profile of lumiracoxib as compared to celecoxib
To assess the efficacy of lumiracoxib as compared to celecoxib with respect to:
Overall OA pain intensity on a 0-100 mm VAS by visit
Patient's global assessment of disease activity by visit
Physician's global assessment of disease activity by visit
Patient's functional status using the WOMAC 3.1 LK sub-scale scores and total score by visit
Usage of rescue medication
Response to treatment according to OARSI criteria by visit

CONTACTS AND LOCATIONS:
Locations (15):
- Novartis Investigative Site, Malvern, Australia
- Novartis Investigative Site, Vienna, Austria
- Novartis Investigative Site, Prague, Czechia
- Novartis Investigative Site, Turku, Finland
- Novartis Investigative Site, Dresden, Germany
- Novartis Investigative Site, Budapest, Hungary
- Novartis Investigative Site, Haifa, Israel
- Novartis Investigative Site, Lisse, Netherlands
- Novartis Investigative Site, Rotorua, New Zealand
- Novartis Investigative Site, Poznan, Poland
- Novartis Investigative Site, Bratislava, Slovakia
- Novartis Investigative Site, Johannesburg, South Africa
- Novartis Investigative Site, Seville, Spain
- Novartis Investigative Site, Uppsala, Sweden
- Novartis Investigative Site, Izmir, Turkey (Türkiye)